CLINICAL TRIAL: NCT00617968
Title: A Multicenter, Randomized, Open-label, Phase II Study to Evaluate the Efficacy and Safety of Neoadjuvant Treatment Consisting of Either a Docetaxel - Letrozole Combination or Letrozole Alone in Women Over 60 Years of Age Suffering From Grade I or II Operable Hormone Receptor-positive Breast Tumor.
Brief Title: GETNA2 Neoadj. TAX+Femara vs Femara in g I/II Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Nathalie Billon/Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976D_2502
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: DOCETAXEL

SUMMARY:
Primarily to evaluate the rates of clinical and radiological response in the 2 groups. Secondarily rate of histological response.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer histologically proven by microbiopsy (14G or 16G) enabling confirmation of the diagnosis, and evaluation of the histological prognostic grade, hormonal receptors and HER2 status.
* Tumor T2 or T3, non-metastasized, non-inflammatory, unilateral
* Clinically or radiologically measurable lesion greater than 2 cm (ultrasound and/or mammogram)
* Receptors RE+ and/or RP+ (positive status determined according to the criteria of the investigating centers)
* HER 2 / neu status of 0, 1+ or 2+ in immunohistochemistry
* Histological grade I or II
* Menopausal patients aged greater than or equal to 60 years
* Patients with ECOG PS greater than or equal to 2
* Satisfactory hematological, hepatic and renal functions:
* Hemoglobin greater than or equal to 10 g/dL
* Platelet count greater than or equal to 100x109/L
* Polynuclear neutrophil count greater than 1.5x109/L
* Creatinine less than or equal to ≤ 1.5 ULN
* AST/ALT less than or equal to 1.5 ULN
* Alkaline phosphatases less than or equal to 2.5 ULN
* Patients able to be followed throughout the study
* Patient's consent obtained.

Exclusion Criteria:

* Inflammatory or T4 breast cancer
* T1 tumor
* Patients whose tumor is deemed by the doctor to be difficult to evaluate
* Tumor that is metastatic from the outset (M1) or locally advanced and inoperable from the outset
* RE and RP receptors negative or unknown
* HER 2/neu positive at 3 +
* Non-menopausal patients
* Surgical biopsy and/or ganglion dissection before neoadjuvant treatment
* Significant poorly controlled cardiac disorders, such as unstable angina pectoris, poorly controlled heart failure, arrhythmia requiring treatment, or myocardial infarction within the last 3 months
* Cardiovascular, hepatic, neurological or endocrine disease, or other major systemic disease that makes it difficult to conduct the protocol or to interpret the results
* Previous history of cancer that occurred within the last 10 years, with the exception of cervical cancers and basocellular skin cancers that were properly treated
* Allergy to polysorbate 80
* Hypersensitivity to docetaxel
* Participation in another clinical trial with one of the study medicinal products during the 30 days prior to entry in the study
* Patients who are unable to undergo medical monitoring for geographical, social or psychological reasons

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-10; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Rate of clinical and radiological response evaluated according to RECIST criteria | During the study conduct

SECONDARY OUTCOMES:
Rate of histological response | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BILLON, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France